CLINICAL TRIAL: NCT02507375
Title: Phase Ib, Open-label, Multi-center Study of the Combination of Pertuzumab and Erlotinib in Patients With Locally Advanced or Metastatic (Stage IIIb/IV) NSCLC After Failure of at Least One Prior Chemotherapy Regimen.
Brief Title: A Study of Pertuzumab With Erlotinib in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO20024; NCT02514096 (obsolete NCT alias)
Record Dates: First submitted 2015-07-14; First posted 2015-07-23 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; pertuzumab

ARMS (2):
- Cohort 1 (Experimental): Participants will receive IV infusion of pertuzumab at a loading dose of 840 mg on Day 1, followed by a dose of 420 mg every 3 weeks. Erlotinib will be administered daily, at a dose level of 100 mg orally (PO).
  Interventions: Drug: Erlotinib; Drug: Pertuzumab
- Cohort 2 (Experimental): Participants will receive IV infusion of pertuzumab at a loading dose of 840 mg on Day 1, followed by a dose of 420 mg every 3 weeks. Erlotinib will be administered daily, at a dose level of 150 mg orally (PO).
  Interventions: Drug: Erlotinib; Drug: Pertuzumab

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be administered as oral tablets.
  Other Names: Tarceva
Drug: Pertuzumab — Pertuzumab will be administered as intravenous (IV) infusion.
  Other Names: Perjeta

SUMMARY:
This study will assess the safety and tolerability, and make a preliminary assessment of activity, of a combination of pertuzumab and erlotinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who have failed on at least one prior chemotherapy regimen. The anticipated time on study treatment is until disease progression or unacceptable toxicity, and the target sample size is less than 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than or equal to 18 years of age
* Histological confirmation of non-small cell lung cancer (NSCLC)
* Locally advanced or metastatic disease
* Failure of at least one prior regimen of standard chemotherapy for locally advanced or metastatic disease
* Life expectancy of more than or equal to 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Baseline Left Ventricular Ejection Fraction (LVEF) of greater than or equal to 50%
* A negative pregnancy test one week prior to treatment and willingness to use contraception among women of childbearing potential
* Availability of histological Formalin-Fixed, Paraffin-Embedded (FFPE) tumor tissue

Exclusion Criteria:

* Prior chemotherapy, radiotherapy or immunotherapy within 4 weeks of study Day -8
* Prior treatment with any agent which targets growth factors or their receptors
* Patients who have not recovered from the acute reversible effects of chemotherapy and radiotherapy
* History of clinically significant cardiovascular disease
* History or evidence of central nervous system metastases
* Treatment with any investigational drug within 28 days of the start of the study (day -8)
* Prior cumulative doxorubicin dose of more than 360 mg/m2 or the equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (3):
- Antwerp, Belgium
- Barcelona, Spain
- Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventeen patients enrolled in 3 centers. Three patients from cohort 1 and 1 patient from cohort 2 completed the 6 cycles of study therapy, as planned.
Pre-assignment Details: Two participants in cohort 2 did not begin experimental study drug treatment in Cycle 1, so were not included in the analysis set.The resulting participant flow includes only participants who received pertuzumab.
Groups:
- Erlotinib 100 mg + Pertuzumab 420 mg: Participants received erlotinib 100 mg orally once daily plus pertuzumab 420 mg intravenously every 3 weeks until disease progression, unacceptable toxicity, or the participant withdrew from the study. The first dose of pertuzumab was a loading dose of 840 mg intravenously
- Erlotinib 150 mg + Pertuzumab 420 mg: Participants received erlotinib 150 mg orally once daily plus pertuzumab 420 mg intravenously every 3 weeks until disease progression, unacceptable toxicity, or the participant withdrew from the study. The first dose of pertuzumab was a loading dose of 840 mg intravenously.
Period: Overall Study
Arm/Group | Erlotinib 100 mg + Pertuzumab 420 mg | Erlotinib 150 mg + Pertuzumab 420 mg
Started | 6 | 9 (Two patients in cohort 2 did not begin treatment in Cycle 1 so were not included in the analysis set)
Cycle 1 | 6 | 9
Received Pertuzumab | 6 | 6
Cycle 2 | 5 | 5
Cycle 3 | 4 | 5
Cycle 4 | 4 | 2
Cycle 5 | 3 | 1
Cycle 6 | 3 | 1
Extension Period | 2 | 1
Completed | 2 | 1
Not Completed | 4 | 8
Not completed — Progressive Disease | 4 | 5
Not completed — Death | 0 | 1
Not completed — Refused treatment | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All recruited participants who received at least 1 dose of both pertuzumab and erlotinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib 100 mg + Pertuzumab 420 mg | Erlotinib 150 mg + Pertuzumab 420 mg | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (5.89) | 56.0 (10.28) | 60.2 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 0 | 1
  United Kingdom | 1 | 1 | 2
  Spain | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as: Any non-hematological toxicity ≥ Grade 3 according to the Common Terminology Criteria for Adverse Events, version 3.0, except for fever, chills, and flu-like symptoms, which occurred despite adequate participant management. The following Grade 1-3 toxicities were exempt: Grade 1-3 skin and/or epithelial toxicities consistent with erlotinib single agent therapy, unless they did not respond to treatment or dose reduction or interruption (Grade 4 skin and/or epithelial toxicities were considered to be a DLT); Grade 4 neutropenia occurring for > 7 days; febrile neutropenia which occurred despite adequate participant management; Grade 4 thrombocytopenia or any thrombocytopenia requiring platelet transfusion; and any subjectively intolerable toxicity felt by the investigator to be related to either one of the compounds.
Time Frame: From baseline to end of the study (up to 42 weeks)
Measure: Number; unit: Percentage of participants
Arm/Group | Erlotinib 100 mg + Pertuzumab 420 mg | Erlotinib 150 mg + Pertuzumab 420 mg
Number analyzed (Participants) | 6 | 6
Percentage of participants | 0 | 0

2. Secondary Outcome: Percentage of Participants Classified as Responders
Description: Responders are participants who achieved either a complete response or a partial response according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria. RECIST is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: within 18 weeks
Population: Full analysis set
Measure: Number; unit: percentage of participants
Groups:
- Total Population: Erlotinib + pertuzumab
Arm/Group | Total Population | Erlotinib 100 mg + Pertuzumab 420 mg | Erlotinib 150 mg + Pertuzumab 420 mg
Number analyzed (Participants) | 15 | 6 | 9
percentage of participants | 20 | 33.3 | 11.1

3. Secondary Outcome: Percentage of Participants With a Complete Response or Partial Response at the End of Cycles 1, 2, 3, 4, and 6
Description: Complete and partial responses were determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. A complete response was defined as the disappearance of all target and non-target lesions. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter.
Time Frame: From baseline to the end of the study (up to 42 weeks)
Measure: Number; unit: Percentage of participants
Arm/Group | Erlotinib 100 mg + Pertuzumab 420 mg | Erlotinib 150 mg + Pertuzumab 420 mg
Number analyzed (Participants) | 6 | 9
Percentage of participants
  Cycle 1 | 0 | 0
  Cycle 2 | 33.3 | 11.1
  Cycle 3 | 0 | 0
  Cycle 4 | 33.3 | 11.1
  Cycle 6 | 16.7 | 11.1

4. Secondary Outcome: Peak Plasma Concentration (Cmax) for Pertuzumab (Cycle 2) in the Presence of Erlotinib (at Steady-state) in Patients With NSCLC
Description: Maximum Observed Plasma Concentration (Cmax), which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered, typically measured in nanograms/milliliter (ng/mL), reported as mg/L.
Time Frame: on day 1 of cycle 2, 1 hour pre-dose and 0.5, 1.5, 4, 8, 24, 168, 336 and 504 hours after the start of the infusion
Population: Pharmacokinetic analysis subset, defined as all participants from either cohort with adequate data for performing PK analysis
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Pertuzumab + Erlotinib: In cycle 1 day 1 pertuzumab was administered at a dose of 840mg over 60 min. All patients included in the pharmacokinetic (PK) analyses of pertuzumab (cycle 2 only), tolerated the infusion in cycle 1 as the cycle 2 dose of 420mg was administered over 30 mins in all but one patient, who was dosed over 33 minutes. Serum samples for pertuzumab were taken for pharmacokinetic analysis on day 1 of cycle 2, 1 hour pre-dose and 0.5, 1.5, 4, 8, 24, 168, 336 and 504 hours after the start of the infusion. Four participants in each cohort (8 total) had adequate data to be included in the PK analyses.
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 8
mg/L | 231 (55.3)

5. Secondary Outcome: Time of Cmax (Tmax) for Pertuzumab (Cycle 2) in the Presence of Erlotinib (at Steady-state) in Patients With NSCLC
Description: The time at which maximum concentration (Cmax), which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered, is reached (Tmax).
Time Frame: on day 1 of cycle 2, 1 hour pre-dose and 0.5, 1.5, 4, 8, 24, 168, 336 and 504 hours after the start of the infusion
Population: PK analysis subset
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 8
days | 0.23 (0.11)

6. Secondary Outcome: Terminal Phase Plasma Half-life (t ½) for Pertuzumab (Cycle 2) in the Presence of Erlotinib (at Steady-state) in Patients With NSCLC
Description: Terminal phase plasma half-life (t ½) is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, rather than the time required to eliminate half the administered dose.
Time Frame: on day 1 of cycle 2, 1 hour pre-dose and 0.5, 1.5, 4, 8, 24, 168, 336 and 504 hours after the start of the infusion
Population: PK analysis subset with adequate data for this analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 6
days | 17.9 (2.18)

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) for Pertuzumab (Cycle 2) in the Presence of Erlotinib (at Steady-state) in Patients With Non-small Cell Lung Cancer (NSCLC)
Description: Bioavailability [AUC(0-t)] is a measure of how much of the drug reaches the person's bloodstream from time 0 (pre-dose) to a given time point (t) for the body to use. The extent of product bioavailability is estimated by the area under the blood concentration vs time curve. The Area Under the Curve (AUC) is calculated by plotting the drug's blood levels on a graph at different times during the set period. The area under this curve reflects the amount of drug exposure in the set time period, calculated as hour * nanograms (ng) per milliliter (mL), which equates to mg.day/L. Bioavailability Extrapolated to Infinity [AUC (0-inf)] is a calculated measure of how much of the drug will ever reach the person's bloodstream for the body to use. AUC (0-inf) stands for the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (forever). It is obtained from calculating AUC (0-t) plus AUC (t-inf).
Time Frame: on day 1 of cycle 2, 1 hour pre-dose and 0.5, 1.5, 4, 8, 24, 168, 336 and 504 hours after the start of the infusion
Population: Pharmacokinetic analysis subset with appropriate data available
Measure: Mean (Standard Deviation); unit: mg*day/L
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 8
mg*day/L
  AUC(0-21 days) n=8 | 1780 (340)
  AUC(0-inf) n=7 | 3000 (815)

8. Secondary Outcome: Clearance (CL) for Pertuzumab (Cycle 2) in the Presence of Erlotinib (at Steady-state) in Patients With NSCLC
Description: A fundamental concept in pharmacokinetics is drug clearance (CL), that is, elimination of drugs from the body. The clearance is simply the ratio of the dose to the area under the curve (AUC), so that the higher the AUC for a given dose, the lower the clearance. If a drug is administered by continuous infusion and a steady state is achieved, the clearance can be estimated from a single measurement of the plasma drug concentration.
Time Frame: on day 1 of cycle 2, 1 hour pre-dose and 0.5, 1.5, 4, 8, 24, 168, 336 and 504 hours after the start of the infusion
Population: PK subset
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 8
L/day | 0.24 (0.05)

9. Secondary Outcome: Volume of Distribution at Steady-state (Vss) for Pertuzumab (Cycle 2) in the Presence of Erlotinib (at Steady-state) in Patients With NSCLC
Description: Steady-state volume of distribution of a drug is an estimate of drug distribution independent of elimination processes. It is most useful for predicting the plasma concentrations following multiple dosing to a steady-state or pseudo-equilibrium. Vss is proportional to the amount of drug in the body versus the plasma concentration of the drug at steady state (pseudo-equilibrium). It is a calculated measure.
Time Frame: on day 1 of cycle 2, 1 hour pre-dose and 0.5, 1.5, 4, 8, 24, 168, 336 and 504 hours after the start of the infusion
Population: PK analysis subset
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 8
Liters | 4.9 (1.3)

ADVERSE EVENTS:
Time Frame: Timeframe was up to 42 weeks
Description: All participants who received at least 1 dose of both pertuzumab and erlotinib and had at least 1 post-baseline safety follow-up.
Groups:
- Cohort 1: Erlotinib 100 mg + pertuzumab 420 mg
- Cohort 2: Erlotinib 150 mg + pertuzumab 420 mg
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 4/9
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=9)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung Cancer Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Sudden death due to progressive disease
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=9)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Nail Bed Inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (3)
Mucosal Inflammation (General disorders) | 1 (1) | 1 (1)
Axillary Pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 1 (1)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Nail Infection (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral Fungal Infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Per Version A the protocol was halted for 2 DLTs (grade 3 manageable rash common for erlotinib) in the first 6 patients. Ethics committee approved redefining DLT and starting anew with Version B. No further DLTs were observed throughout the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study.

The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.